CLINICAL TRIAL: NCT00008411
Title: Phase III Study Comparing the Use of Docetaxel on a Every Three-Week vs. Weekly Schedule in the Treatment of Patients With Metastatic Breast Cancer
Brief Title: Docetaxel in Treating Patients With Metastatic Breast Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ID99-242; P30CA016672 (NIH); MDA-ID-99242 (Other: UT MD Anderson Cancer Center); AVENTIS-MDA-ID-99242; NCI-1691; CDR0000068408 (Registry Identifier: NCI PDQ)
Record Dates: First submitted 2001-01-06; First posted 2003-01-27 (Estimated); Last update posted 2012-07-30 (Estimated); Status verified 2012-07

CONDITIONS: Breast Cancer
Keywords: stage IV breast cancer; recurrent breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Docetaxel Weekly (Experimental): Arm I: Docetaxel IV over 1 hour on day 1. Courses repeat every 21 days.
  Interventions: Drug: Docetaxel
- Docetaxel Every 3 Weeks (Experimental): Arm II: Docetaxel IV over 30 minutes on days 1, 8, and 15. Courses repeat every 28 days.
  Interventions: Drug: Docetaxel

INTERVENTIONS:
Drug: Docetaxel — Every 3 weeks at a starting dose of 75 mg/m2 IV over 1 hour on day 1, repeated every 21 days.
  Other Names: Taxotere
  Arms: Docetaxel Every 3 Weeks
Drug: Docetaxel — 35 mg/m2 IV over 30 minutes on days 1, 8, and 15, for 3 weeks followed by one week of rest repeated every 28 days.
  Other Names: Taxotere
  Arms: Docetaxel Weekly

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Randomized phase III trial to determine the effectiveness of docetaxel in treating patients who have metastatic breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the objective tumor response rate, duration of response, time to progression, progression-free survival, and overall survival in women with metastatic breast cancer treated with docetaxel administered weekly vs every three weeks.
* Compare the safety and toxicity of these regimens in these patients.
* Evaluate the maintenance of relative dose intensity with each regimen in these patients.
* Correlate pretreatment serum HER2/neu level and response with docetaxel therapy in these patients.

OUTLINE: This is a randomized, multicenter study. Patients are stratified according to prior taxane use (yes vs no), number of prior chemotherapy regimens for metastatic disease (0 vs 1), and participating center. Patients are randomized to one of two treatment arms.

* Arm I: Patients receive docetaxel IV over 1 hour on day 1. Courses repeat every 21 days.
* Arm II: Patients receive docetaxel IV over 30 minutes on days 1, 8, and 15. Courses repeat every 28 days.

Treatment continues in both arms in the absence of disease progression or unacceptable toxicity.

Patients are followed at 3 weeks, at 3, 6, 9, and 12 months, and then annually for 4 years.

PROJECTED ACCRUAL: A total of 160 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed metastatic breast cancer
* Bidimensionally measurable disease
* No uncontrolled brain metastases or leptomeningeal disease
* Hormone receptor status:

  * Not specified

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Sex:

* Female

Menopausal status:

* Not specified

Performance status:

* Zubrod 0-2

Life expectancy:

* At least 3 months

Hematopoietic:

* Platelet count at least 100,000/mm^3
* Neutrophil count at least 1,000/mm^3
* Hemoglobin at least 8 g/dL

Hepatic:

* Bilirubin no greater than upper limit of normal (ULN)
* SGOT/SGPT no greater than 1.5 times ULN (2.5 times ULN provided alkaline phosphatase no greater than ULN)
* Alkaline phosphatase no greater than 2.5 times ULN (4 times ULN provided transaminases no greater than ULN)

Renal:

* Creatinine no greater than 2.0 mg/dL

Neurologic:

* No peripheral neuropathy grade 2 or greater
* Neurologic status must be stable 2 weeks after surgery and/or radiotherapy for brain metastasis
* No psychiatric disorders

Other:

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No other malignancy within the past 5 years except non-melanoma skin cancer, carcinoma in situ of the cervix, or other curatively treated malignancy
* No other serious condition or illness, including active infection
* No history of hypersensitivity to polysorbate 80

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* Recovered from prior chemotherapy
* No more than 2 prior chemotherapy regimens (no more than 1 prior regimen for metastatic disease)
* No prior paclitaxel or docetaxel (except in the adjuvant setting)
* At least 12 months since prior adjuvant taxane (paclitaxel or docetaxel)
* Prior anthracycline-based therapy allowed

Endocrine therapy:

* Not specified

Radiotherapy:

* At least 2 weeks since prior radiotherapy and recovered

Surgery:

* At least 2 weeks since prior surgery and recovered

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 1999-12; Primary Completion 2006-03 (Actual); Study Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
Objective Tumor Response Rate | Weekly

CONTACTS AND LOCATIONS:
Overall Officials: Edgardo Rivera, MD, Study Chair — M.D. Anderson Cancer Center
Locations (2):
- United States (2):
  - MD Anderson Cancer Center at University of Texas, Houston, Texas
  - University of Texas M.D. Anderson CCOP Research Base, Houston, Texas

REFERENCES:
- [Result] Rivera E, Mejia JA, Arun BK, Adinin RB, Walters RS, Brewster A, Broglio KR, Yin G, Esmaeli B, Hortobagyi GN, Valero V. Phase 3 study comparing the use of docetaxel on an every-3-week versus weekly schedule in the treatment of metastatic breast cancer. Cancer. 2008 Apr 1;112(7):1455-61. doi: 10.1002/cncr.23321. PMID 18300256
- See also: UT MD Anderson Cancer Center Website — http://www.mdanderson.org